CLINICAL TRIAL: NCT02241096
Title: Pharmacokinetics of Intravenous Lidocaine Infusion in Children
Brief Title: PK Intravenous Lidocaine Infusion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of available study participants.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-3194
Record Dates: First submitted 2014-09-04; First posted 2014-09-16 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lidocaine (Experimental): IV lidocaine bolus of 1.5mg/kg over 10 minutes followed by a 1mg/kg/hr IV lidocaine infusion.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — IV lidocaine bolus of 1.5mg/kg over 10 minutes followed by a 1mg/kg/hr IV lidocaine infusion.
  Other Names: xylocaine

SUMMARY:
To determine safe concentration level of lidocaine infusion in children.

DETAILED DESCRIPTION:
This study will address the working hypothesis that intravenous lidocaine may be administered as a bolus followed by an infusion with reliable and safe blood levels of lidocaine. Serial blood draws will be obtained to determine safety of lidocaine doses used in this study by measuring blood levels of lidocaine and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* male or female children 3-15 years of age
* ASA physical status 1-3
* scheduled for colorectal surgery with abdominal incision

Exclusion Criteria:

* ASA physical status > 3
* postoperative intubation planned ahead of surgery
* history of chronic use of opioid (use longer than 3 months)
* history of hepatic, renal, or cardiac failure
* history of significant liver disease including liver failure, acute or chronic hepatitis, hepatomegaly, portal hypertension and elevated liver enzymes
* history of organ transplant
* BMI > 30
* history of cardiac arrhythmia
* history of long QT syndrome
* history of allergic reaction to lidocaine or similar agents
* history of seizure disorder
* patient without PICC or other central access with contraindication to inhalation induction
* family history or known patient susceptibility to malignant hyperthermia

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safe serum levels of lidocaine infusion (<5 mcg/ml of lidocaine in blood) | Samples will be collected until the end of the OR case and up to 24 hours after surgery
  Blood samples will be obtained at predetermined times after start and finish of lidocaine infusion. Each sample is 1ml. Samples will be obtained at the baseline placement of IV, 0 - 3 minutes after bolus has completed, 9 - 15 minutes after bolus infusion, 4 minutes prior to end or at the end of the continuous infusion, 55 - 65 following the end of infusion, 2 - 7 hours after completion of continuous infusion and 20 - 24 hours after completion of infusion if clinical labs are also necessary.

SECONDARY OUTCOMES:
Safe metabolite levels (monoethylglycinexylidide (MEGX) and glycinexylidide (GX) with intraoperative IV lidocaine infusions | Samples will be collected until the end of the OR case and up to 24 hours after surgery
  We will monitor monoethylglycinexylidide (MEGX) and glycinexylidide (GX).
  Blood samples (1ml each) for metabolites will be as follows: baseline with initial placement, 4 minutes after infusion completed, 2 - 7 hours after infusion completion, 20 - 24 hours after infusion completion if clinical labs are being drawn

CONTACTS AND LOCATIONS:
Overall Officials: Smokey J Clay, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Candiotti KA, Yang Z, Morris R, Yang J, Crescimone NA, Sanchez GC, Bird V, Leveillee R, Rodriguez Y, Liu H, Zhang YD, Bethea JR, Gitlin MC. Polymorphism in the interleukin-1 receptor antagonist gene is associated with serum interleukin-1 receptor antagonist concentrations and postoperative opioid consumption. Anesthesiology. 2011 May;114(5):1162-8. doi: 10.1097/ALN.0b013e318216e9cb. PMID 21455057
- [Background] Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesth Analg. 2009 Nov;109(5):1464-9. doi: 10.1213/ANE.0b013e3181bab1bd. PMID 19843784
- [Background] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Background] Harvey KP, Adair JD, Isho M, Robinson R. Can intravenous lidocaine decrease postsurgical ileus and shorten hospital stay in elective bowel surgery? A pilot study and literature review. Am J Surg. 2009 Aug;198(2):231-6. doi: 10.1016/j.amjsurg.2008.10.015. Epub 2009 Mar 12. PMID 19285304
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307